CLINICAL TRIAL: NCT00815451
Title: Effect of Polyphenols on Glucoregulatory Biomarkers, Blood Pressure and Lipid Profile in Overweight and Obese Subjects
Brief Title: Effect of Polyphenol-rich Dark Chocolate on Obesity
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Queen Margaret University (Other)
Responsible Party: suzana almoosawi, PhD student QMU
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: 1-salmoosawi
Record Dates: First submitted 2008-12-29; First posted 2008-12-30 (Estimated); Last update posted 2009-09-18 (Estimated); Status verified 2009-09

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- placebo dark chocolate (Placebo Comparator): polyphenol-poor dark chocolate
  Interventions: Dietary Supplement: placebo
- polyphenol-rich dark chocolate (Experimental)
  Interventions: Dietary Supplement: Acticoa polyphenol-rich dark chocolate

INTERVENTIONS:
Dietary Supplement: placebo — polyphenol-free dark chocolate 20g to be distributed throughout the day for 4 weeks
  Other Names: barry callebaut
  Arms: placebo dark chocolate
Dietary Supplement: Acticoa polyphenol-rich dark chocolate — 20g to be distributed throughout the day for 4 weeks
  Other Names: barry callebaut, acticoa
  Arms: polyphenol-rich dark chocolate

SUMMARY:
This study aims to investigate the effect of polyphenol-rich dark chocolate (DC) on insulin resistance, adiponectin , blood pressure (BP), lipid profile in obese subjects and determine possible associations between all assessed parameters.

It hypothesizes that consumption of polyphenol-rich Dc could lower fasting glucose levels, insulin resistance and improve BP, total cholesterol, low-density lipoprotein (LDL) and triglycerides while increasing adiponectin and high-density lipoprotein (HDL) in overweight or obese individuals.

DETAILED DESCRIPTION:
It is well acknowledged that the main mechanism by which cocoa and DC polyphenols improve fasting glucose levels, insulin sensitivity, BP and lipid profile in healthy individuals and those with hypertension and/or impaired glucose-tolerance, involves increased nitric oxide (NO) bioavailability. NO is essential for the regulation of blood pressure, glucose and lipid balance. This is evident in that e-NOsynthase knockout mice exhibit insulin resistance, hypertension and hyperlipidemia, a cluster of diseases that is also observed in the metabolic syndrome. Recently, it was shown that adiponectin regulates eNOsynthase activity through the phosphatidylinositol 3-kinase-dependent pathway wherein eNOsynthase is phosphorylated by 5'-AMP-activated protein kinase at Ser1179 and that plasma adiponectin levels are inversely correlated with BMI, waist-to-hip ratio, fasting plasma glucose, insulin, triglyceride, hyperinsulinemia, and glucose intolerance and positively with HDL-cholesterol, but not BP. This suggests a strong link between impaired NO bioavailability, adiponectin levels and obesity. Indeed, apart from exhibiting impaired NO bioavailability, obese individuals also have decreased plasma adiponectin levels. Since cocoa and DC are known to modulate NO activity, investigating the impact of cocoa or DC polyphenols on adiponectin levels and observing a correlation between its levels and improved fasting glucose levels, insulin resistance, BP and lipid profile is essential in improving our understanding of the relationship between diet and health, particularly that polyphenols in apples, oolong and green tea polyphenols have been previously shown to influence adiponectin levels.

This study uses a randomised single-blind, placebo-controlled design. Following a 1-week run-in phase, each group will be randomised to one of the two groups: placebo-polyphenol-rich DC, polyphenol-rich DC-placebo. Subjects will follow each diet for 4weeks, after which they will cross-over to the next diet separated by a 2-week washout period and until each subject completes both interventions.

ELIGIBILITY:
Inclusion Criteria:

* Healthy female volunteers
* Aged 18-50 years
* Group 1 will consist of volunteers with BMI of 18-25 kg/m2
* Group 2 will consist of women with BMI of 25-35 kg/m2

Exclusion Criteria:

* Cardiovascular disease
* Hypertension
* Diabetes
* Smokers
* People taking dietary supplements
* Hypertension or cholesterol-lowering drugs
* Those with high cocoa or DC intake, soy or nut allergies

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2008-11; Primary Completion 2009-10 (Estimated); Study Completion 2009-12 (Estimated)

PRIMARY OUTCOMES:
adiponectin | week 0, 4, 6, 10

SECONDARY OUTCOMES:
insulin sensitivity | week 0, 4, 6, 10
blood pressure | week 0, 4, 6, 10
lipid profile | week 0, 4, 6, 10

CONTACTS AND LOCATIONS:
Overall Officials: suzana h almoosawi, BScHons HN, Principal Investigator — QMU
Locations (1):
- Queen margaret university, Musselburgh, east lothian, United Kingdom